CLINICAL TRIAL: NCT03761264
Title: Clinical, Microbiological and Quality of Life Outcomes Following Use of Systemic and Local Antimicrobials in the Management of Odontogenic Infections in Paediatric Patients
Brief Title: Systemic and Local Antimicrobials in the Management of Dental Abscess in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Shani Ann Mani, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP053A-17HTM
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Dentoalveolar Abscess
Keywords: Odontogenic Infections; Paediatric Patients; Local Antimicrobials; Systemic Antimicrobials; Dentoalveolar Abscess; Apical Dentoalveolar Abscess; Periapical Abscess; Suppurative Periapical Periodontitis
MeSH Terms: conditions — Periapical Abscess | interventions — Pulpdent; Amoxicillin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Intra-canal Odontopaste® (Experimental): Single visit placement of Odontopaste®
  Interventions: Drug: Odontopaste®
- Intra-canal Pulpdent (Active Comparator): Single visit placement of Pulpdent
  Interventions: Drug: Pulpdent
- Oral Amoxicillin (Active Comparator): Amoxicillin 15mg/kg tds for 5 days
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Odontopaste® — Teeth with abscess will be opened from the crown to allow cleaning of the canals following which the Odontopaste® will be placed in the canals and the pulp chamber. Cavity will be sealed with capsulated Glass ionomer cement.
  Other Names: Zinc Oxide based endodontic dressing
  Arms: Intra-canal Odontopaste®
Drug: Pulpdent — Teeth with abscess will be opened from the crown to allow cleaning of the canals following which the Pulpdent paste will be placed in the canals and the pulp chamber. Cavity will be sealed with capsulated Glass ionomer cement.
  Other Names: Calcium hydroxide endodontic paste
  Arms: Intra-canal Pulpdent
Drug: Amoxicillin — Teeth with abscess will be opened from the crown to allow cleaning of the canals . A sterile cotton pellet will be placed in the pulp chamber and cavity sealed with capsulated Glass ionomer cement. The patient will be prescribed oral amoxicillin at 15mg/kg body weight tds for 5 days
  Other Names: Amoxycillin
  Arms: Oral Amoxicillin

SUMMARY:
Dental infections originating in the teeth are routinely managed systemically with a course of oral antibiotics, while severe forms are managed with intravenous antibiotics. Dental infections can also be managed by removing the offending cause of the infection followed by placement of an intra-canal medication which acts as a local antimicrobial. Intra-canal medicaments are being used in clinical practice following root canal treatment. The investigators hypothesize that the effect of intra-canal antimicrobials in the management of dental infections will be the better than oral antibiotics in terms of clinical , microbial and oral- health quality of life parameters. This will be a three-arm, parallel, comparative, randomized study with the aim of assessing the efficacy of intra-canal medication and oral antibiotics in reducing the infection and treatment of odontogenic infections, based on signs and symptoms and microbial count. The study will be performed in child participants between the age group of 3 to 11 years presenting with acute odontogenic infections. Participants will be randomized by block randomization. The treatment duration of the study will be at least 5 days or maximum 7 days depending upon the response. Participants will be assessed on Day 3 and Day 5/7. Concurrently, the oral health-related quality of life (OHRQoL) following these clinical interventions in children will be recorded and again on Day 14. Quantitative assessment of microorganisms seen in the root canals and the changes seen in the microbial flora through the treatment will help us to determine the best antimicrobial agent to be used in the management of odontogenic infections.

DETAILED DESCRIPTION:
This study will comprise of a three-arm, parallel, comparative, randomized treatment of children aged 3 to 11 years presenting with acute odontogenic infection. The three arms of the study includes 1) Odontopaste® as a one time intra-canal placement, 2) Calcium hydroxide (gold standard) as a one time intra-canal placement and 3) a course of amoxicillin three times daily for 5 days administered orally with meal. Patients will not receive additional medical therapy such as analgesics or anti-inflammatory drugs. The participants will be selected for the treatment based on a block randomization in groups of three. On Day 1 after confirming the eligibility based on clinical examination and radiographic finding, informed consent will be obtained. At baseline (Day 1), clinical parameters including pain,swelling, regional lymphadenitis, percussion of the tooth, trismus, fistula and pus discharge will be recorded. Participant will undergo an intervention whereby the tooth will be opened from the clinical crown followed by microbiological sampling, drainage and irrigation of the tooth, intra-canal medicament placed in the canals according to randomization and the cavity sealed with a Glass ionomer cement. Participants in the oral antibiotic group will have no intra-canal medicament placed and instead a sterile cotton pellet placed. Simultaneously, the Malay-ECOHIS will be given to the parent/guardian of the participant. The microbiological sampling will be stored in an appropriate transport medium and sent to the central laboratory for quantitative assessment via quantitative polymerase chain reaction (qPCR) using SYBR® Green. Participants will be assessed on Day 3 for clinical parameters and the integrity of restoration. The next and final assessment will be done at Day 5/7, where clinical parameters will be recorded along with microbiological sampling as in Day 1. The Malay-ECOHIS survey will be repeated. The primary objective of the study is to assess the resolution of the infection based on 1) clinical parameters, 2) microbiological sampling and 3) oral health quality of life. The treatment will be carried out by five operators who are calibrated and the individual sub components such as recording clinical parameters, microbiological sampling and assessing the OHRQoL questionnaire will be carried out by the same operator respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with acute odontogenic infections on primary teeth with evidence of intra-oral / extra- oral swelling and pus discharge
* Absence of any systemic disease
* Age group between 3-11 years
* Malaysian citizen

Exclusion Criteria:

* Patients taking antibiotics 30 days prior to their attendance to the department
* Presence of any systemic disease
* Patients with cellulitis
* Patients suffering from spreading odontogenic infections which require hospitalization or immediate IV antibiotic treatment
* Tooth with poor prognosis for extraction
* Extensively resorbed roots (> 2/3rd)
* Patients allergic or resistance to amoxicillin
* Non-Malaysian citizen

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Mean Change From Baseline in Wong Baker Faces Pain Rating Scale of Pain Score at Day 3, Day 5 or 7 | Baseline, Days 3, 5 or 7
  Wong Baker Faces Pain Rating Scale (WBFPRS) is used to measure the amount of pain that a participant experiences. This scale has numerical ratings from 0 to 10. Zero indicates no pain and 10 indicates worst possible pain. Change in Pain is documented as WBFPRS score at Baseline and subsequent reviews.
Mean Change From Baseline in Visual Rating Scale of Swelling Score at Days 3, 5 or 7 | Baseline, Days 3, 5 or 7
  Visual Rating Scale (VRS) is used to measure the degree of swelling that the participant experiences. This scale has numerical ratings from 0 to 5. Zero indicates no swelling pain and 5 indicates worse swelling imaginable. Change in Swelling is documented as VRS score at Baseline and subsequent reviews.
Mean Change From Baseline in Regional Lymphadenitis Score at Days 3, 5 or 7 | Baseline, Days 3, 5 or 7
  Examination of lymph nodes is performed and recorded as 0,1 and 2. Zero indicates no inflammation of lymph nodes; 1 is described as inflammation of regional lymph nodes, palpatory examination painless, and a score of 2 indicates inflammation of regional lymph nodes, palpatory examination painful.
Mean Change From Baseline in Temperature Score at Days 3, 5 or 7 | Baseline, Days 3, 5 or 7
  Temperature is recorded as baseline and on review visits as 0,1 and 2. Zero indicates afebrile (up to 36.9 °C),1 as subfebrile (37-37.9 °C) and 2 as febrile (38 °C and more)
Mean Change From Baseline in Trismus Score at Days 3, 5 or 7 | Baseline, Days 3, 5 or 7
  Distance measurement between incisal ridge of upper and lower jaw in case a patient had the teeth and in case the teeth were missing the measurement was based on the distance between alveolar ridges of the frontal region. The measured results were evaluated according to the established scale: 0 - there is no trismus (21 mm and more),1 - slightly pronounce trismus (11- 20 mm) and score 2 as very pronounced trismus (0 -10 mm).
Mean Change From Baseline in Percussion Score at Days 3, 5 or 7 | Baseline, Days 3, 5 or 7
  Percussion is performed as light tapping on the tooth using the edge of a mouth mirror and recorded as 0 and 1. Zero is recorded as no tenderness and 1 as presence of tenderness.
Mean Change From Baseline in Fistula Score at Days 3, 5 or 7 | Baseline, Days 3, 5 or 7
  Fistula is examined clinically and recorded as 0 and 1. Zero is recorded as absence of fistula and 1 as presence of fistula
Mean Change From Baseline in Pus Discharge Score at Days 3, 5 or 7 | Baseline, Days 3, 5 or 7
  Clinical examination on the abscessed tooth to document pus discharge as 0 and 1. Zero is recorded as no pus discharge and 1 as presence of pus discharge.
Mean Reduction in Bacterial Count by quantitative Polymerase Chain Reaction (q-PCR) From Baseline and at Day 5 or 7 | Baseline, Day 5 or Day 7
  Quantitative assesment by q-PCR using SYBR® Green will show the count of oral anaerobes on Day 1 and Day 5 or 7 of treatment.
Mean change of ECOHIS scores from baseline and at Day 5 or Day 7 | Baseline, Day 5 or Day 7
  Malay-ECOHIS comprises of child impact section and family impact section. Under child impact section consist of 4 domains which are symptom, function,psychology and self image and social interaction. Whilst, under family impact section consist of 2 domains which are parental distress and family function. Each question has six response options: 0=never; 1 = hardly ever; 2 = sometimes; 3 = often; 4 = very often; and 5 = "I don't know". The results will show differences in ECOHIS scores between the modes of treatments from baseline and at Day 5 or Day 7.

SECONDARY OUTCOMES:
Quantification of Individual Target Species | First 2 Months of Study
  A particular species of the most common bacteria seen in the root canal will be identified using meta-genomic analysis and the five most commonly seen bacteria will be chosen as target species.

CONTACTS AND LOCATIONS:
Overall Officials: Shani Ann Mani Dr, Principal Investigator — Department of Paediatric Dentistry, Faculty of Dentistry, University of Malaya; Syarida Hasnur Dr, Principal Investigator — Department of Restorative Dentistry, Faculty of Dentistry, University of Malaya; Lily Azura Shoaib Dr, Principal Investigator — Department of Paediatric Dentistry, Faculty of Dentistry, University of Malaya
Locations (1):
- University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Caufield PW, Griffen AL. Dental caries. An infectious and transmissible disease. Pediatr Clin North Am. 2000 Oct;47(5):1001-19, v. doi: 10.1016/s0031-3955(05)70255-8. PMID 11059347
- [Background] Nair PN. Pathogenesis of apical periodontitis and the causes of endodontic failures. Crit Rev Oral Biol Med. 2004 Nov 1;15(6):348-81. doi: 10.1177/154411130401500604. PMID 15574679
- [Background] Robertson D, Smith AJ. The microbiology of the acute dental abscess. J Med Microbiol. 2009 Feb;58(Pt 2):155-162. doi: 10.1099/jmm.0.003517-0. PMID 19141730
- [Background] Walsh LJ. Serious complications of endodontic infections: some cautionary tales. Aust Dent J. 1997 Jun;42(3):156-9. doi: 10.1111/j.1834-7819.1997.tb00113.x. PMID 9241924
- [Background] Fouad AF, Rivera EM, Walton RE. Penicillin as a supplement in resolving the localized acute apical abscess. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1996 May;81(5):590-5. doi: 10.1016/s1079-2104(96)80054-0. PMID 8734709
- [Background] Lewis MA. Why we must reduce dental prescription of antibiotics: European Union Antibiotic Awareness Day. Br Dent J. 2008 Nov 22;205(10):537-8. doi: 10.1038/sj.bdj.2008.984. PMID 19023306
- [Background] Dar-Odeh N, Ryalat S, Shayyab M, Abu-Hammad O. Analysis of clinical records of dental patients attending Jordan University Hospital: Documentation of drug prescriptions and local anesthetic injections. Ther Clin Risk Manag. 2008 Oct;4(5):1111-7. doi: 10.2147/tcrm.s3727. PMID 19209291
- [Background] Dar-Odeh NS, Abu-Hammad OA, Al-Omiri MK, Khraisat AS, Shehabi AA. Antibiotic prescribing practices by dentists: a review. Ther Clin Risk Manag. 2010 Jul 21;6:301-6. doi: 10.2147/tcrm.s9736. PMID 20668712
- [Background] Hills-Smith H, Schuman NJ. Antibiotic therapy in pediatric dentistry. II. Treatment of oral infection and management of systemic disease. Pediatr Dent. 1983 Mar;5(1):45-50. No abstract available. PMID 6344030
- [Background] Bansal R, Jain A. Overview on the current antibiotic containing agents used in endodontics. N Am J Med Sci. 2014 Aug;6(8):351-8. doi: 10.4103/1947-2714.139277. PMID 25210667
- [Background] Farhad A, Mohammadi Z. Calcium hydroxide: a review. Int Dent J. 2005 Oct;55(5):293-301. doi: 10.1111/j.1875-595x.2005.tb00326.x. PMID 16245464
- [Background] Rodd HD, Waterhouse PJ, Fuks AB, Fayle SA, Moffat MA; British Society of Paediatric Dentistry. Pulp therapy for primary molars. Int J Paediatr Dent. 2006 Sep;16 Suppl 1:15-23. doi: 10.1111/j.1365-263X.2006.00774.x. No abstract available. PMID 16939452
- [Background] Matijevic S, Lazic Z, Kuljic-Kapulica N, Nonkovic Z. Empirical antimicrobial therapy of acute dentoalveolar abscess. Vojnosanit Pregl. 2009 Jul;66(7):544-50. doi: 10.2298/vsp0907544m. PMID 19678579
- [Background] Novaes TF, Pontes LRA, Freitas JG, Acosta CP, Andrade KCE, Guedes RS, Ardenghi TM, Imparato JCP, Braga MM, Raggio DP, Mendes FM; CARDEC collaborative group. Responsiveness of the Early Childhood Oral Health Impact Scale (ECOHIS) is related to dental treatment complexity. Health Qual Life Outcomes. 2017 Sep 20;15(1):182. doi: 10.1186/s12955-017-0756-z. PMID 28931398
- [Background] Siqueira JF Jr, Rocas IN, Lopes HP. Patterns of microbial colonization in primary root canal infections. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2002 Feb;93(2):174-8. doi: 10.1067/moe.2002.119910. PMID 11862207
- [Background] Frisch MB, Clark MP, Rouse SV, Rudd MD, Paweleck JK, Greenstone A, Kopplin DA. Predictive and treatment validity of life satisfaction and the quality of life inventory. Assessment. 2005 Mar;12(1):66-78. doi: 10.1177/1073191104268006. PMID 15695744
- [Background] Locker D. Measuring oral health: a conceptual framework. Community Dent Health. 1988 Mar;5(1):3-18. No abstract available. PMID 3285972
- [Background] Jackson SL, Vann WF Jr, Kotch JB, Pahel BT, Lee JY. Impact of poor oral health on children's school attendance and performance. Am J Public Health. 2011 Oct;101(10):1900-6. doi: 10.2105/AJPH.2010.200915. Epub 2011 Feb 17. PMID 21330579
- [Background] Al-Malik M, Al-Sarheed M. Pattern of management of oro-facial infection in children: A retrospective. Saudi J Biol Sci. 2017 Sep;24(6):1375-1379. doi: 10.1016/j.sjbs.2016.03.004. Epub 2016 Mar 31. PMID 28855834
- See also: Intra Canal Treatments for Clinical Success and Patient Comfort — http://pdfs.semanticscholar.org/2e49/67ff2f0a06e4b4707d3f0b1436d7b437d91f.pdf
- See also: American Association of Endodontics (AAE) Guidance on the Use of Systemic Antibiotics in Endodontics — http://www.aae.org/specialty/wp-content/uploads/sites/2/2017/06/aae_systemic-antibiotics.pdf
- See also: The early childhood oral health impact scale (ECOHIS): Assessment tool in oral health related quality of life — http://www.researchgate.net/publication/325111490_The_early_childhood_oral_health_impact_scale_ECOHIS_Assessment_tool_in_oral_health_related_quality_of_life
- See also: Bacteriology of Infected Deciduous Root Canal -A Review — http://www.researchgate.net/publication/277103677_Bacteriology_of_infected_deciduous_root_canal_a_review

DOCUMENTS (2):
  • Study Protocol (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT03761264/Prot_000.pdf
  • Informed Consent Form (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT03761264/ICF_001.pdf